CLINICAL TRIAL: NCT07004140
Title: Proving Utility of a New Field-cycling MRI Prototype in Acute Stroke Patients
Acronym: PUFFINS 3
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2-001-25; 25/SS/0021 (Other: NHS Scotland A Research Ethics Committee)
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Stroke Acute
Keywords: Stroke; Field-Cycling Imaging; FCI
MeSH Terms: conditions — Stroke | interventions — Blood Specimen Collection; In Vitro Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ischaemic stroke: Ischaemic stroke patients within 24 hours from symptom onset
  Interventions: Other: 3T MRI research scan; Other: Field-Cycling Imaging research scan; Other: Follow up 3T MRI research scan; Other: Follow up Field-Cycling Imaging research scan; Other: Blood samples for clotting experiments in vitro
- Haemorrhagic stroke: Patients with primary intracerebral haemorrhage within 24 hours from symptom onset
  Interventions: Other: 3T MRI research scan; Other: Field-Cycling Imaging research scan

INTERVENTIONS:
Other: 3T MRI research scan — Baseline MRI scan
Other: Field-Cycling Imaging research scan — Baseline FCI scan
Other: Follow up 3T MRI research scan — Day 30 3T MRI scan
  Groups: Ischaemic stroke
Other: Follow up Field-Cycling Imaging research scan — Day 30 FCI scan
  Groups: Ischaemic stroke
Other: Blood samples for clotting experiments in vitro — Thrombi from whole blood from ischaemic stroke patients will be formed and examined using bench top nuclear magnetic resonance (NMR) assays. At baseline and 30 days after stroke onset.
  Groups: Ischaemic stroke

SUMMARY:
The goal of this study is to test if a new type of MRI scanner, called Field-Cycling Imaging (FCI), can show changes in the brain within the first day of a stroke due to a blocked blood vessel or bleeding in the brain. The main question it aims to answer is:

• Can FCI identify brain tissue that might recover within the first few hours after a stroke begins?

Participants will undergo a standard MRI scan and an FCI scan, as soon as possible after hospital admission.

Participants who have had a blocked blood vessel will also provide a blood sample and will have a follow up visit at 30 days for repeat of both scans and providing another blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke (<24 hours from symptom onset).
* NIHSS ≥4 and <25 with cortical involvement and/or large vessel occlusion on baseline imaging.
* Able to undergo 3T and FCI MRI <24h of onset.
* With or without thrombolysis.

Exclusion Criteria:

* Contraindications to MRI.
* Medically unstable.
* Unable to comprehend or comply with instructions regarding scanning
* Prior mRS of >3.
* Identified for thrombectomy.
* Non-stroke pathology or previous cortical infarct on CT scan > 1/3 of middle cerebral artery territory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with acute stroke admitted to Aberdeen Royal Infirmary.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Agreement between extent of ischaemic stroke at-risk tissue/infarct core obtained from FCI dispersion maps and 3T MRI modalities at baseline | Baseline at stroke onset
  Receiver operator curves (ROC) curves comparing extent of at-risk tissue/infarct core obtained from FCI dispersion maps and from 3T MRI modalities at baseline at stroke onset.

SECONDARY OUTCOMES:
Agreement between extent of haemorrhagic volume obtained from FCI dispersion maps and 3T MRI modalities at baseline | Baseline at stroke onset
  Receiver operator curves (ROC) curves comparing extent of haemorrhagic volume obtained from FCI dispersion maps and from 3T MRI modalities at baseline at stroke onset.
Agreement of infarct core volume measurements obtained from FCI and 3T MRI at day 30 in ischaemic stroke patients | 30 days after stroke onset
  Comparison of infarct core volumes on 30-day 3T FLAIR and baseline/30-day FCI T1 dispersion maps in ischaemic stroke patients.
Agreement between T1 dispersion curve measurements obtained from in vivo clot in large intracerebral vessels and clot formed in vitro. | At baseline and 30 days after stroke onset
  Extent of agreement between quantified T1 dispersion curve measurements obtained from in vivo imaging and benchtop Fast Field Cycling Nuclear Magnetic Resonance (FFC-NMR). Extent of correlation between thrombo-elastography measurements against in vivo measurements of T1 dispersion.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mallikourti V, Ross PJ, Maier O, Guzman-Gutierrez G, Franko E, Lurie DJ, Broche LM, Macleod MJ. Field-Cycling MRI for Identifying Minor Ischemic Stroke Below 0.2 T. Radiology. 2024 Aug;312(2):e232972. doi: 10.1148/radiol.232972. PMID 39189899
- [Background] Senn N, Ross PJ, Ayde R, Mallikourti V, Krishna A, James C, de Vries CF, Broche LM, Waiter GD, MacLeod MJ. Field-cycling imaging yields repeatable brain R1 dispersion measurement at fields strengths below 0.2 Tesla with optimal fitting routine. MAGMA. 2025 Jul;38(3):465-474. doi: 10.1007/s10334-025-01230-w. Epub 2025 Feb 15. PMID 39955477